CLINICAL TRIAL: NCT04135872
Title: Relationship Between Baseline Serum Albumin Level and Cognitive Impariment in Mild Acute Ischemic Stroke
Brief Title: Hypoalbuminemia in Mild Acute Stroke and Cognitive Impariment Post-stroke
Status: Completed | Type: Observational
Sponsor: Dongguan People's Hospital (Other Government)
Responsible Party: Principal Investigator, Zhu Shi, Deputy Director of Neurology, Dongguan People's Hospital
Other Study IDs: DongguanPeopleHospital
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Cognitive Impairment; Stroke; Albumin; Double
MeSH Terms: conditions — Cognitive Dysfunction; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — fasting venous blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypoalbuminemia: hypoalbuminemia was classified as serum albumin level (SAL) <35g/L
  Interventions: Other: strengthened nuitritional treatment
- normal albumin level: patients with serum albumin level (SAL) of 35g/L or higher

INTERVENTIONS:
Other: strengthened nuitritional treatment — improving nutritional status by nasal feeding for dysphagia or iv. albumin when serum albumin level lower than 35g/L
  Groups: hypoalbuminemia

SUMMARY:
This registration enrolled patients with acute ischemic stroke within 72 hours after stroke ictus. Patients was identified as first-ever stroke based on past medical histrory. Admission CT was conducted to exclude hemorrhagic stroke, but not those bleeding transformation after ischemia injury. Baseline characteristics, including demographics, vascular risk factors, lab tests and neuroimagings were collected. Patients were followed up for cognitive assessments.

DETAILED DESCRIPTION:
This is a perspective stroke registry cohort study. Stroke patients were included if ：(1) acute first-ever ischemic stroke and admitted within 72 hours after onset; (2) clinical stroke diagnosis was confirmed with positive diffusion-weighted magnetic resonance imaging (DW-MRI), those with isolated posterior circulations infarcts were exclude ; (3) presented with mild stroke severity ( admission NIHSS score ≤5); (4) age between 40 and 80 years.

Clinical data including demographic characteristics, risk factors, and baseline NIHSS score were assessed and collected using a standardized table by experienced neurologists. Lab tests were performed with fasting venous blood samples within 18 hours of admission.

Patients were followed up for 6 months. The cognitive functions were assessed using the Chinese version of Montreal Cognitive Assessment (MoCA).

Contributing factors to post-stroke cognitive impariment (PSCI) were determined by comparing clinical data between PSCI and non-PSCI groups. All potential confounders were introduced into the multivariate regression models.

ELIGIBILITY:
Inclusion Criteria:

1. acute first-ever ischemic stroke and admitted within 72 hours after onset;
2. clinical stroke diagnosis was confirmed with positive diffusion-weighted magnetic resonance imaging (DW-MRI), those with isolated posterior circulations infarcts were exclude ;
3. presented with mild stroke severity ( admission NIHSS score ≤5);
4. age between 40 and 80 years.

Exclusion Criteria:

1. Patients with index cognitive impairment or under current anti-dementia or psychiatric medication;
2. patients with large infarcts (≥1/3 middle cerebral artery territory);
3. patients with severe language or physical disability that impede neuropsychological testing;
4. patients with recurrent transient ischemic attack (TIA)/stroke during follow-up;
5. coexisting serious conditions known to impair cognitive function

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients were continuously enrolled from a perspective stroke registry between January 1, 2017 and June 31, 2018, in Dongguan People's Hospital, Guangdong, China.
Sampling Method: Non-Probability Sample
Enrollment: 435 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
PSCI | 6 months post-stroke
  Patients with a MoCA score of <24 were categorized as having PSCI

CONTACTS AND LOCATIONS:
Overall Officials: zhu shi, Principal Investigator — dongguan peoples hospital
Locations (1):
- Dongguan Peoples' Hospital, Dongguan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
The final decision to release IPD is still pending because of the ongoing census among all paticipants's decision.